CLINICAL TRIAL: NCT03041116
Title: Efficacy, Safety, and Tolerability of Fosmetpantotenate (RE-024), a Phosphopantothenate Replacement Therapy, in Pantothenate Kinase-Associated Neurodegeneration (PKAN) Patients: A Randomized, Double-Blind, Placebo-Controlled Study With an Open-Label Extension
Brief Title: Efficacy and Safety Study of Fosmetpantotenate (RE-024) in PKAN Participants
Acronym: PKAN
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was terminated since fosmetpantotenate did not show statistically significant effects or clinical benefits during the double-blind period.
Sponsor: Travere Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 024PKAN15004
Record Dates: First submitted 2016-12-02; First posted 2017-02-02 (Estimated); Results first posted 2020-12-29 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Pantothenate Kinase-Associated Neurodegeneration
Keywords: PKAN
MeSH Terms: conditions — Pantothenate Kinase-Associated Neurodegeneration | interventions — fosmetpantotenate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Fosmetpantotenate (Experimental): Administered as powder for reconstitution.
  Interventions: Drug: Fosmetpantotenate
- Placebo (Placebo Comparator): Administered as powder for reconstitution.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fosmetpantotenate — Daily dosing
  Other Names: RE-024
  Arms: Fosmetpantotenate
Drug: Placebo — Daily dosing
  Arms: Placebo

SUMMARY:
This study investigated whether fosmetpantotenate (RE-024), a phosphopantothenate replacement therapy, was safe and effective in treating participants with PKAN.

ELIGIBILITY:
Inclusion Criteria:

1. The participant had a diagnosis of PKAN as indicated by confirmed mutations in the pantothenate kinase 2 gene.
2. The participant was male or female aged 6 to 65 years, inclusive.
3. The participant had a score of ≥ 6 on the PKAN-specific activities of daily living measure.

Exclusion Criteria:

1. The participant had required regular or intermittent invasive ventilatory support to maintain vital signs within 24 weeks prior to randomization.
2. The participant had a deep brain stimulation device implanted within 6 months prior to screening.
3. The participant had taken deferiprone within 30 days prior to screening.
4. The participant was unable to maintain stable doses of allowed concomitant medications for the first 24 weeks of the study.

Ages: 6 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2017-07-17 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Klopstock, MD, Principal Investigator — Klinikum der Universität München
Locations (19):
- United States (9):
  - Travere Investigational Site, Irvine, California
  - Travere Investigational Site, Washington D.C., District of Columbia
  - Travere Investigational Site, Miami, Florida
  - Travere Investigational Site, Decatur, Georgia
  - Travere Investigational Site, Chicago, Illinois
  - Travere Investigational Site, Boston, Massachusetts
  - Travere Investigational Site, New York, New York
  - Travere Investigational Site, Pittsburgh, Pennsylvania
  - Travere Investigational Site, Houston, Texas
- Travere Investigational Site, Toronto, Ontario, Canada
- Travere Investigational Site, Prague, NAP, Czechia
- France (2):
  - Travere Investigational Site, Montpellier, Languedoc-Rousillon
  - Travere Investigational Site, Paris, Île-de-France Region
- Travere Investigational Site, München, Bavaria, Germany
- Travere Investigational Site, Milan, Italy
- Travere Investigational Site, Oslo, Norway
- Travere Investigational Site, Warsaw, Poland
- Spain (2):
  - Travere Investigational Site, Barcelona, Catalonia
  - Travere Investigational Site, Barcelona

REFERENCES:
- [Result] Klopstock T, Escolar ML, Marshall RD, Perez-Duenas B, Tuller S, Videnovic A, Greblikas F. The FOsmetpantotenate Replacement Therapy (FORT) randomized, double-blind, Placebo-controlled pivotal trial: Study design and development methodology of a novel primary efficacy outcome in patients with pantothenate kinase-associated neurodegeneration. Clin Trials. 2019 Aug;16(4):410-418. doi: 10.1177/1740774519845673. Epub 2019 May 6. PMID 31055958

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in Spain, United States, Canada, Czech Republic, France, Germany, Italy, Norway, and Poland from 17-July-2017 to 23-December-2019. A total of 91 participants were screened, of which 84 participants were randomized in the double blind period, and 78 participants completed the double-blind period.
Pre-assignment Details: The study consisted of a screening period of up to 29 days. All assessments at screening were done as per the schedule of assessments.
Groups:
- Fosmetpantotenate: Double-blind Period: each randomized participant received an oral dose of fosmetpantotenate with dose escalation for Days 1 through 3, followed by the full dose 3 times daily (TID) from Day 4, based on the participant's age and weight at screening, for 24 weeks.
  Open-label Period: all participants continued treatment with fosmetpantotenate according to the dose they were receiving at the end of the double-blind period. No dose escalation was required.
- Placebo: Double-blind Period: each randomized participant received an oral dose of placebo matched to fosmetpantotenate with dose escalation for Days 1 through 3, followed by the full dose TID from Day 4, based on the participant's age and weight at screening, for 24 weeks.
  Open-label Period: all participants started treatment with fosmetpantotenate according to the placebo dose they were receiving at the end of the double-blind period. No dose escalation was required.
Period: Double-blind
Arm/Group | Fosmetpantotenate | Placebo
Started | 41 | 43
Received at Least 1 Dose of Study Drug | 41 | 43
Completed | 41 | 37
Not Completed | 0 | 6
Not completed — Death | 0 | 2
Not completed — Withdrawal by Subject | 0 | 4
Period: Open-label
Arm/Group | Fosmetpantotenate | Placebo
Started | 41 | 37
Received At Least 1 Dose of Study Drug | 41 | 37
Completed | 0 | 0
Not Completed | 41 | 37
Not completed — Death | 1 | 0
Not completed — Termination of the study by Sponsor | 39 | 37
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population: any participant who received at least 1 dose of study drug during any period of the study.
Groups:
- Fosmetpantotenate: Double-blind Period: each randomized participant received an oral dose of fosmetpantotenate with dose escalation for Days 1 through 3, followed by the full dose TID from Day 4, based on the participant's age and weight at screening, for 24 weeks.
  Open-label Period: all participants continued treatment with fosmetpantotenate according to the dose they were receiving at the end of the double-blind period. No dose escalation was required.
- Total: Total of all reporting groups
Arm/Group | Fosmetpantotenate | Placebo | Total
Number analyzed (Participants) | 41 | 43 | 84
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.6 (10.61) | 23.1 (13.56) | 22.9 (12.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 19 | 39
  Male | 21 | 24 | 45
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 2 | 10
  Not Hispanic or Latino | 28 | 36 | 64
  Unknown or Not Reported | 5 | 5 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 4 | 4
  White | 25 | 28 | 53
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 13 | 9 | 22

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline In The Pantothenate Kinase-Associated Neurodegeneration-Activities of Daily Living (PKAN-ADL) Total Score To The End Of The 24-week Double-blind Period
Description: Change from baseline to Week 24 activities of daily living was assessed on the PKAN-ADL scale based on the Unified Parkinson's Disease Rating Scale (UPDRS) Part II. The PKAN-ADL is a validated measure of the participant's ability to complete ADL that are impacted by the diffuse motor manifestations of PKAN. It consists of 12 items related to activities of daily living, including eating, dressing, and walking. Each item has responses ranging from 0-4, with a higher value indicating greater disability in the given activity. To compute the total score, responses are summed across the 12 items. The available range of total scores on the PKAN-ADL scale was from 0 (no ADL affected) to 48 (ADL highly affected). The reported least square mean (LSM) was adjusted for baseline score and age group from the Type III analysis. A decrease in score indicates improvement in symptoms.
Time Frame: Baseline (Day -1), Week 24
Population: Double-blind Full Analysis Set: any participant who received at least 1 dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Fosmetpantotenate | Placebo
Number analyzed (Participants) | 41 | 43
units on a scale | -1.3 (0.56) | -1.3 (0.58)
Statistical Analysis 1: Comparison: Fosmetpantotenate vs Placebo; Test type: Superiority; p = 0.9115, Mixed Models Analysis — p-value was derived from test of contrast between treatment effects using LSM estimate, adjusted for baseline score and age group from Type III analysis. The test of contrast at Week 24 was considered the primary comparison; Difference in LS Mean = -0.1, 95% CI 2-sided [-1.69 to 1.51], Standard Error of Mean 0.8

2. Primary Outcome: Number Of Participants With At Least 1 (≥1) Treatment-emergent Adverse Event (TEAE) And Treatment-emergent Serious Adverse Event (TESAE) During The 24-week Double-blind Period
Description: An adverse event (AE) is any untoward medical occurrence associated with the use of the investigational product (IP; active or placebo) in a participant, without regard to possibility of causal relationship with IP. A serious adverse event (SAE) is an AE resulting in any of the following outcomes: death; initial or prolonged inpatient hospitalization; life threatening experience (immediate risk of death from AE); persistent or significant disability/incapacity; congenital anomaly/birth defect; other medically important serious medical events. The TEAEs in the double-blind period are defined as AEs that are new or are a worsening of an existing condition that begins from day of first dose of IP until day after last dose for double-blind treatment period.
Time Frame: From Screening until end of Week 24
Population: Safety Population: any participant who received at least 1 dose of study drug during any period of the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Fosmetpantotenate | Placebo
Number analyzed (Participants) | 41 | 43
Participants
  ≥1 TEAE | 34 | 35
  ≥1 TESAE | 8 | 6

3. Secondary Outcome: Absolute Change From Baseline In The UPDRS Part 3 (UPDRS-III) Total Score To The End Of The 24-week Double-blind Period
Description: The UPDRS is a comprehensive assessment of the burden and severity of signs and symptoms of Parkinsonism captured via systematic interview and neurological examination. The UPDRS-III is a standardized neurological examination that evaluates the performance of movements commonly affected in Parkinson's disease, PKAN, and other movement disorders. Part III of the UPDRS consists of 27 items, which correspond to 14 domains related to motor abilities such as tremor, stability, and bradykinesia. Each item has responses ranging from 0-4. To compute the UPDRS-III total score, responses are summed across the 27 items, and accordingly, range from 0-108. For domain totals, responses are summed across all of the items in a given domain (when domain corresponds to multiple items). An increase in score indicates greater disability. The reported LSM was adjusted for baseline score and age group from the Type III analysis.
Time Frame: Baseline (Day -1), Week 24
Population: Double-blind Full Analysis Set: any participant who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fosmetpantotenate | Placebo
Number analyzed (Participants) | 41 | 43
units on a scale | 0.7 (5.25) | -1.0 (6.81)
Statistical Analysis 1: Comparison: Fosmetpantotenate vs Placebo; Test type: Superiority; p = 0.1421, Mixed Models Analysis — p-value was derived from the test of contrast between treatment effects using the LSM estimate, adjusted for baseline score and age group from the Type III analysis. The test of contrast at week 24 was considered the primary comparison; Difference in LS Mean = 2, 95% CI 2-sided [-0.7 to 4.78], Standard Error of Mean 1.38

ADVERSE EVENTS:
Time Frame: From Screening until end of treatment (approximately 29 Months)
Description: The TEAEs in the double-blind period were defined as AEs that were new or a worsening of an existing condition that began from the day of the first dose of IP until the day after the last dose for the double-blind treatment period. The TEAEs in the open-label period were defined as AEs that were new or a worsening of an existing condition that began from the day of the first dose of IP received during the open-label period until 30 days after last dose for the open-label period.
Groups:
- Fosmetpantotenate: Double-blind Period: each randomized participant received an oral dose of fosmetpantotenate with dose escalation for Days 1 through 3, followed by the full dose TID from Day 4, based on the participant's age and weight at screening, for 24 weeks.
  Open-label Period: all participants continued treatment with fosmetpantotenate according to the dose they were receiving at the end of the double-blind period. No dose escalation was required.
  Includes data over the entire study for those who completed the double-blind period and entered the open-label period.
- Placebo: Double-blind Period: each randomized participant received an oral dose of placebo matched to fosmetpantotenate with dose escalation for Days 1 through 3, followed by the full dose TID from Day 4, based on the participant's age and weight at screening, for 24 weeks.
  Open-label Period: all participants started treatment with fosmetpantotenate according to the placebo dose they were receiving at the end of the double-blind period. No dose escalation was required.
  Includes data over the entire study for those who completed the double-blind period and entered the open-label period.
- Fosmetpantotenate During Double-blind Period: Double-blind Period: each randomized participant received oral dose of fosmetpantotenate with dose escalation for Days 1 through 3, followed by the full dose TID from Day 4, based on the participant's age and weight at screening, for 24 weeks.
- Placebo During Double-blind Period: Double-blind Period: each randomized participant received oral dose of placebo matched to fosmetpantotenate with dose escalation for Days 1 through 3, followed by the full dose TID from Day 4, based on the participant's age and weight at screening, for 24 weeks.
- Fosmetpantotenate During Open-label Period: Open-label Period: at Week 25, all participants continued treatment with fosmetpantotenate according to the dose they were receiving at the end of the double-blind period. No dose escalation was required.
- Placebo During Open-label Period: Open-label Period: at Week 25, all participants started treatment with fosmetpantotenate according to the placebo-matched dose they were receiving at the end of the double-blind period. No dose escalation was required.
Arm/Group | Fosmetpantotenate | Placebo | Fosmetpantotenate During Double-blind Period | Placebo During Double-blind Period | Fosmetpantotenate During Open-label Period | Placebo During Open-label Period
All-Cause Mortality (participants affected / at risk) | 1/41 | 2/37 | 0/41 | 2/43 | 1/41 | 0/37
Serious Adverse Events (participants affected / at risk) | 9/41 | 9/37 | 8/41 | 6/43 | 4/41 | 9/37
Other Adverse Events (participants affected / at risk) | 35/41 | 25/37 | 34/41 | 35/43 | 25/41 | 26/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fosmetpantotenate (N=41) | Placebo (N=37) | Fosmetpantotenate During Double-blind Period (N=41) | Placebo During Double-blind Period (N=43) | Fosmetpantotenate During Open-label Period (N=41) | Placebo During Open-label Period (N=37)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Shunt malfunction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fracture treatment (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dystonia (Nervous system disorders) | 4 (6) | 4 (5) | 2 (3) | 1 (1) | 2 (3) | 4 (5)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Multiple sclerosis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Generalised tonic-clonic seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotonia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nervous system disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Disease progression (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Faecaloma (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin Infections (Infections and infestations) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinovirus infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis streptococcal (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fosmetpantotenate (N=41) | Placebo (N=37) | Fosmetpantotenate During Double-blind Period (N=41) | Placebo During Double-blind Period (N=43) | Fosmetpantotenate During Open-label Period (N=41) | Placebo During Open-label Period (N=37)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 7 (8) | 1 (1) | 5 (6) | 4 (4) | 2 (2) | 1 (1)
Discomfort (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Feeling cold (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
General physical health deterioration (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Generalised oedema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Medical device site inflammation (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Medical device site rash (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Sleep disorder (Psychiatric disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Adjustment disorder with depressed mood (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Restlessness (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Affect lability (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrostomy tube site complication (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0) | 2 (4) | 1 (1) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Face injury (Injury, poisoning and procedural complications) | 1 (2) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Foetal exposure during pregnancy (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Traumatic haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Animal scratch (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eyelid contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Scar (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Traumatic fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 4 (4) | 1 (1) | 4 (4) | 2 (4) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 3 (3) | 0 (0) | 1 (2) | 1 (1) | 3 (3)
Weight decreased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Haemoglobin decreased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Bacterial test positive (Investigations) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Blood cholesterol increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood glucose decreased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac murmur (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coagulation time prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Crystal urine present (Investigations) | 1 (1) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0)
Culture throat positive (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemoglobin urine present (Investigations) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Monocyte count increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Monocyte percentage increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nitrite urine present (Investigations) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Platelet count increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urine leukocyte esterase positive (Investigations) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
White blood cell count decreased (Investigations) | 1 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
White blood cell count increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood urea increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cortisol decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
White blood cells urine positive (Investigations) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Prothrombin time prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Urine leukocyte esterase (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Left ventricular hypertrophy (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchial secretion retention (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Choking (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dystonia (Nervous system disorders) | 7 (11) | 3 (3) | 6 (10) | 8 (9) | 1 (1) | 3 (3)
Headache (Nervous system disorders) | 4 (4) | 3 (3) | 2 (2) | 5 (9) | 2 (2) | 3 (3)
Oromandibular dystonia (Nervous system disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1) | 2 (3) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Drooling (Nervous system disorders) | 1 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Dyskinesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle spasticity (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nystagmus (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Multiple sclerosis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nerve compression (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Opisthotonus (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Parkinsonism (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperkinesia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dark circles under eyes (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eczema eyelids (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Optic atrophy (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Visual acuity reduced (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 8 (11) | 2 (2) | 5 (5) | 4 (6) | 3 (6) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 5 (5) | 1 (1) | 4 (4) | 0 (0) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 8 (12) | 2 (2) | 4 (8) | 5 (6) | 4 (4) | 2 (2)
Constipation (Gastrointestinal disorders) | 4 (5) | 2 (2) | 3 (3) | 2 (2) | 2 (2) | 2 (2)
Nausea (Gastrointestinal disorders) | 4 (4) | 0 (0) | 2 (2) | 7 (13) | 2 (2) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1) | 2 (3) | 1 (1) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Faecaloma (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Faeces soft (Gastrointestinal disorders) | 1 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperchlorhydria (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Parotid gland enlargement (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Salivary hypersecretion (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Tongue disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal hypermotility (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Chromaturia (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urine odour abnormal (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (4) | 0 (0) | 1 (3) | 0 (0) | 1 (1) | 0 (0)
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Rash generalised (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Product taste abnormal (Product Issues) | 2 (2) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Device failure (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Device occlusion (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Knee deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Posture abnormal (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Secondary adrenocortical insufficiency (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 3 (3) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 3 (4) | 1 (1) | 3 (4) | 0 (0) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 5 (7) | 1 (1) | 3 (4) | 2 (2) | 2 (3) | 1 (1)
Urinary tract infection (Infections and infestations) | 6 (6) | 2 (2) | 1 (1) | 0 (0) | 5 (5) | 2 (2)
Bronchitis (Infections and infestations) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Genital candidiasis (Infections and infestations) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Skin infection (Infections and infestations) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Helminthic infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Stoma site infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia influenzal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Ear lobe infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was terminated since fosmetpantotenate did not show statistically significant effects or clinical benefits during the double-blind period.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Institution and Investigator agree that because the study is part of a multi-center study, any publication by the Institution/Investigator of the study results shall not be made before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2019-05-23): https://cdn.clinicaltrials.gov/large-docs/16/NCT03041116/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-22): https://cdn.clinicaltrials.gov/large-docs/16/NCT03041116/SAP_001.pdf